CLINICAL TRIAL: NCT01084694
Title: The Impact of Hematopoeitic Stem Cell Transplantation on Primary Caregiver Level of Burden and Distress
Brief Title: Caregiver Burden and Distress in Hematopoeitic Stem Cell Transplant
Status: Completed | Type: Observational
Sponsor: Northside Hospital, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: NSH 888
Record Dates: First submitted 2010-03-09; First posted 2010-03-10 (Estimated); Results first posted 2019-12-03 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Depression; Anxiety; Fatigue; Distress
Keywords: HSCT; Caregiver; Caregiver Burden; Allogeneic Transplant; Autologous Transplant; Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Depression; Anxiety Disorders; Fatigue; Caregiver Burden

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to examine the impact that serving as a caregiver for a patient undergoing hematopoietic stem cell transplant has on the caregiver. This will include looking at the caregiver's level of burden, depression, anxiety, somatic symptoms, fatigue and overall distress. It will also look at whether caregiver burden leads to an increase in hospitalization and overall outcome.

ELIGIBILITY:
Inclusion Criteria:

Patient:

* Any patient undergoing autologous or allogeneic HSCT at The Blood and Marrow Transplant Program at Northside Hospital
* Patients must have a single primary caregiver
* Patients must be willing to comply with all assessments as outlined in the protocol
* Patients must be willing to sign informed consent

Caregiver:

* Must be the primary caregiver for an autologous or allogenic HSCT patient at the Blood and Marrow Transplant Program at Northside Hospital
* Caregiver must be willing to comply will all assessments as outlined in the protocol
* Caregiver must be willing to sign consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be an autologous patient and their caregiver and an allogeneic patient and their caregiver
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-04-19 (Actual); Primary Completion 2017-09-29 (Actual); Study Completion 2018-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Speckhart, PhD, Principal Investigator — Northside Hospital
Locations (1):
- Northside Hospital, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients will be selected from our Program and will be undergoing evaluation for stem cell transplant.
Pre-assignment Details: Patients and caregivers were enrolled as dyads. Data was collected from both patients and caregivers.
Groups:
- Patients Undergoing Autologous Transplant: 50% of patients enrolled in this study will be undergoing autologous transplant with one primary caregiver.
- Patients Undergoing Allogeneic Transplant: 50% of patients enrolled in this study will be undergoing allogeneic transplant with one primary caregiver.
Period: Overall Study
Arm/Group | Patients Undergoing Autologous Transplant | Patients Undergoing Allogeneic Transplant
Started | 50 | 50
Completed | 44 | 30
Not Completed | 6 | 20
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Death | 2 | 12
Not completed — eligibility not maintained | 2 | 7

BASELINE CHARACTERISTICS:
Groups:
- Autologous Transplant: 50 pairs of autologous patients and their caregivers were enrolled
- Allogeneic Transplant: 50 pairs of allogeneic patients and their caregivers were enrolled
- Total: Total of all reporting groups
Arm/Group | Autologous Transplant | Allogeneic Transplant | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants] — Population: 2 autologous caregivers and 4 allogeneic caregivers did not complete their age on the demographics page. Total autologous included = 48. Total allogeneic included = 46
  Participants
    Patients: <=18 years | 0 | 0 | 0
    Patients: Between 18 and 65 years | 35 | 41 | 76
    Patients: >=65 years | 15 | 9 | 24
    Caregivers: number analyzed (Participants) | 48 | 46 | 94
    Caregivers: <=18 years | 0 | 0 | 0
    Caregivers: Between 18 and 65 years | 32 | 34 | 66
    Caregivers: >=65 years | 16 | 12 | 28
Sex: Female, Male [Count of Participants; unit: Participants]
  Patients: Female | 37 | 36 | 73
  Patients: Male | 13 | 14 | 27
  Caregivers: Female | 36 | 36 | 72
  Caregivers: Male | 14 | 14 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Patients: Hispanic or Latino | 0 | 0 | 0
  Patients: Not Hispanic or Latino | 50 | 49 | 99
  Patients: Unknown or Not Reported | 0 | 1 | 1
  Caregivers: Hispanic or Latino | 0 | 0 | 0
  Caregivers: Not Hispanic or Latino | 48 | 47 | 95
  Caregivers: Unknown or Not Reported | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Patients: American Indian or Alaska Native | 0 | 0 | 0
  Patients: Asian | 1 | 0 | 1
  Patients: Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Patients: Black or African American | 12 | 7 | 19
  Patients: White | 37 | 42 | 79
  Patients: More than one race | 0 | 0 | 0
  Patients: Unknown or Not Reported | 0 | 0 | 0
  Caregivers: American Indian or Alaska Native | 0 | 0 | 0
  Caregivers: Asian | 1 | 0 | 1
  Caregivers: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Caregivers: Black or African American | 13 | 6 | 19
  Caregivers: White | 34 | 41 | 75
  Caregivers: More than one race | 0 | 1 | 1
  Caregivers: Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants] — Region of enrollment for patients
  participants
    United States | 50 | 50 | 100
Region of Enrollment [Number; unit: participants] — Region of enrollment for caregivers
  participants
    United States | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Brief Symptom Inventory and Burden Interview
Description: Brief Symptom Inventory (BSI) measures overall distress. Scores can range from 0-72 with the higher score representing a higher level of distress. Each question is 0-4 with 4 being higher levels of distress. Clinically significant level of distress is 25+. Burden Interview is scored on a continuum. No clinically range, but higher scores mean higher feelings of burden. Scores range from 0-88.
  Time frame: BSI scores and Burden scores were compared in caregivers of HSCT patients at preBMT and post BMT (30 days and 1 year).
Time Frame: Baseline, Day 30 & 1 year
Population: 74 caregivers met criteria for analysis
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Autologous Transplant Recipients: patients receiving autologous transplant
- Allogeneic Transplant Recipients: patients receiving allogeneic transplants
Arm/Group | Autologous Transplant Recipients | Allogeneic Transplant Recipients
Number analyzed (Participants) | 44 | 30
units on a scale
  Baseline BSI | 6.2 [0 to 32] | 6.1 [0 to 32]
  Day 30 BSI | 6 [0 to 34] | 5.9 [0 to 32]
  1 year BSI | 5.3 [0 to 39] | 5.2 [0 to 39]
  Baseline Burden | 13.4 [0 to 39] | 13.1 [0 to 39]
  Day 30 Burden | 18.1 [0 to 36] | 17.9 [0 to 35]
  1 year Burden | 18 [0 to 37] | 18 [0 to 36]

2. Secondary Outcome: Patient Distress, Fatigue & Pain Scores
Description: BSI scale 0-72 with the higher score representing higher distress Brief Fatigue inventory 0-90 with the higher score representing higher fatigue Brief Pain inventory 0-120 with the higher score representing higher pain
Time Frame: Baseline, Day 30 & 1 year
Population: This measure was assessed in patients.
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Autologous Transplant Recipients: patients receiving an autologous transplant
- Allogeneic Transplant Recipients: Patients receiving an allogeneic transplant
Arm/Group | Autologous Transplant Recipients | Allogeneic Transplant Recipients
Number analyzed (Participants) | 44 | 30
units on a scale
  Baseline BSI | 9.1 [0 to 30] | 8.9 [0 to 31]
  Baseline BFI | 24 [0 to 59] | 24 [0 to 59]
  Baseline BPI | 15 [0 to 66] | 15 [0 to 66]
  Day 30 BSI | 9.2 [0 to 31] | 9.1 [0 to 32]
  Day 30 BFI | 27 [0 to 66] | 28 [0 to 67]
  Day 30 BPI | 19 [0 to 71] | 19 [0 to 72]
  1 year BSI | 7.8 [0 to 33] | 7.6 [0 to 33]
  1 year BFI | 21 [0 to 63] | 22 [0 to 64]
  1 year BPI | 14 [0 to 70] | 14 [0 to 73]

3. Secondary Outcome: Overall Patient Survival
Description: Number of patients who are alive at 1 year
Time Frame: Pre-transplant to 1 year post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Autologous Transplant Recipients | Allogeneic Transplant Recipients
Number analyzed (Participants) | 50 | 50
Participants | 42 | 38

4. Secondary Outcome: Common Characteristics of Caregivers
Description: 12 demographic characteristics were collected. If common characteristics were found then it would have been analyzed for correlation with caregiver burden and distress
Time Frame: Baseline
Population: Caregivers were analyzed
Measure: Number; unit: common characteristics
Groups:
- Caregivers for Autologous Transplant Recipients: Caregivers of patients who had autologous transplants
- Caregivers for Allogeneic Transplant Recipients: Caregivers for patients who were receiving an allogeneic transplant
Arm/Group | Caregivers for Autologous Transplant Recipients | Caregivers for Allogeneic Transplant Recipients
Number analyzed (Participants) | 50 | 50
common characteristics | 0 | 0

5. Secondary Outcome: Length of Patient Hospitalization
Time Frame: pretransplant to 1 year post-transplant
Measure: Mean (Full Range); unit: days
Arm/Group | Autologous Transplant Recipients | Allogeneic Transplant Recipients
Number analyzed (Participants) | 44 | 30
days | 10.72 [1 to 76] | 29.34 [2 to 119]

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Patients Undergoing Autologous Transplant: Patients undergoing autologous transplant
- Patients Undergoing Allogeneic Transplant: Patients undergoing allogeneic transplant
- Caregivers for Patients Undergoing Autologous Transplant: Caregivers for patients undergoing autologous transplant. Only emotional distress was monitored for the caregivers.
- Caregivers for Patients Undergoing Allogeneic Transplants: Caregivers for patients undergoing allogeneic transplant. Only emotional distress was monitored for the caregivers
Arm/Group | Patients Undergoing Autologous Transplant | Patients Undergoing Allogeneic Transplant | Caregivers for Patients Undergoing Autologous Transplant | Caregivers for Patients Undergoing Allogeneic Transplants
All-Cause Mortality (participants affected / at risk) | 8/50 | 12/50 | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-16): https://cdn.clinicaltrials.gov/large-docs/94/NCT01084694/Prot_SAP_000.pdf